CLINICAL TRIAL: NCT00298467
Title: An Open-label, Fixed-dose, Multicenter, Phase II Study of MDX-060 in Patients With Relapsed or Refractory Classic Systemic or Primary Cutaneous Anaplastic Large Cell Lymphoma
Brief Title: MDX-060 in Patients With Relapsed or Refractory Classic Systemic or Primary Cutaneous Anaplastic Large Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDX060-04
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Lymphoma, Large-Cell
Keywords: ALCL; csALCL; pcALCL; Lymphoma; Non-Hodgkin's Lymphoma; Anaplastic Large Cell Lymphoma; classic systemci Anaplastic Large Cell Lymphoma (csALCL); primary cutaneous Anaplastic Large Cell Lymphoma (pcALCL)
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Primary Cutaneous Anaplastic Large Cell | interventions — iratumumab

INTERVENTIONS:
Drug: MDX-060

SUMMARY:
This study is an open-label, fixed-dose, multicenter study of MDX-060 in patients with ALCL who have relapsed or refractory disease. There will be 3 phases of this study: Induction, Maintenance, and Follow-up. Patients will be required to attend all protocol-required visits in the 4-week Induction Phase, in which administration of MDX-060 will occur, as well as other testing. Patients who complete the Induction Phase may be eligible for additional MDX-060 treatment ever 2 months for 1 year in the Maintenance Phase. Patients who complete the Maintenance Phase with a response of stable disease or better will be followed every 2 months for 1 year or until disease progression. The purpose of this study is to determine objective response rate at Day 50 in patients with relapsed or refractory classic systemic ALCL or primary cutaneous ALCL treated with MDX-060. Other objectives will be evaluated.

DETAILED DESCRIPTION:
This study is an open-label, fixed-dose, multicenter study of MDX-060 in patients with ALCL who have relapsed or refractory disease. There will be 3 phases of this study: Induction, Maintenance, and Follow-up. Patients will be required to attend all protocol-required visits in the 4-week Induction Phase, in which administration of MDX-060 will occur, as well as other testing. Patients who complete the Induction Phase may be eligible for additional MDX-060 treatment ever 2 months for 1 year in the Maintenance Phase. Patients who complete the Maintenance Phase with a response of stable disease or better will be followed every 2 months for 1 year or until disease progression.

The primary objective of the study is to determine the objective response rate (ORR) at Day 50 in patients with relapsed or refractory classic systemic anaplastic large cell lymphoma (csALCL) or primary cutaneous ALCL (pcALCL) treated with MDX-060. The ORR will be based on an adaption of the NCI Response Criteria for Non-Hodgkin's Lymphoma (NHL) for patients with csALCL and will be based on the Physician's Global Assessment (PGA) for patient with pcALCL.

Secondary objectives include 1) characterizing progression-free survival (PFS); 2) determining response duration (RD); 3) characterizing the effect of MDX-060 on health-related Quality of Life (QoL); 4) evaluating patients with pcALCL using an adaption of the NCI Response Criteria for NHL; 5) characterizing the immunogenicity of MDX-060; 6) characterizing the safety of MDX-060; and 7) determining the best objective response rate (BORR) during the Maintenance Phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* confirmed diagnosis of ALCL
* patient with csALCL must be confirmed CD30+
* patients with csALCL must have failed or relapsed following second line (i.e. salvage) chemotherapy or relapsed or failed following autologous stem cell transplant.
* patients with pcALCL must have progressed after treatment with local radiation therapy or surgical excision or failed systemic therapy with a single agent or multi-agent regimen.
* patients with pcALCL must be confirmed CD30+
* ECOG performance of 0 to 2
* at least 12 years of age
* life expectancy 12 weeks or greater
* must meet screening laboratory values
* women must be post-menopausal for at least 1 year; surgically incapable of bearing children; or utilizing a reliable form of contraception. All women must have a negative pregnancy test.
* men must agree to the use of male contraception for the duration of the study
* patients on corticosteroids must be tapered off the medication 2 weeks prior to the first MDX-060 administration and remain off corticosteroids until day 365.

Exclusion Criteria:

* previous treatment with any anti-CD30 antibody
* history of allogenic transplantation
* any tumor lesion 10 cm or greater in diameter
* any other malignancy, excluding basal or squamous cell carcinoma of the skin, or cervical carcinoma in situ. Any cancer from which the patient has been disease free for at least 5 years is permissible.
* any significant acter or chronic infection.
* prior known serum positivity for HIV, hepatitis B or C as determined at screening.
* treatment with an investigational agent within 30 days or 5 half-lives (whichever is longer) of study screening.
* apparent active or latent tuberculosis infection (TB).
* patients who are pregnant or nursing
* any underlying medical condition which, in the investigator's opinion, will make the administration of MDX-060 hazardous or obscure the interpretation of adverse events.
* concomitant chemotherapy, corticosteroids, investigational agents, other anti-ALCL biologics, or radiation therapy
* patients with mycosis fungoides, or
* patients with recurrent, self-healing papulonodular eruptions only or any other lymphoma other than ALCL.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-02

PRIMARY OUTCOMES:
Objective response rate
progression free survival
response duration
Quality of Life
Immunogenicity
best objective response rate
safety

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - City of Hope, National Medical Center, Duarte, California
  - California Oncology of the Central Valley, Fresno, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Mayo Clinic, Rochester, Minnesota
  - The Cancer Institute of New Jersey - Robert Wood Johnson Unv. Hosp., New Brunswick, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
- Centre Hospitalier Regional Unv. de Lille, Hopital Claude Huriez, Lille, France